CLINICAL TRIAL: NCT00742469
Title: A Randomized,Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Rifaximin for the Prevention of Travellers' Diarrhea
Brief Title: Rifaximin for Prevention of Travellers' Diarrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RFID3003
Record Dates: First submitted 2008-08-24; First posted 2008-08-27 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Diarrhea
Keywords: TD; traveller's diarrhea; campylobacter; shigella; salmonella; E. coli; diarrhea
MeSH Terms: conditions — Diarrhea; Dysentery, Bacillary; Escherichia coli Infections | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Rifaximin
  Interventions: Drug: Rifaximin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine if 600 mg of rifaximin, taken once a day for 14 days by healthy subjects, is safe and effective for the prevention of travellers' diarrhea compared to placebo.

DETAILED DESCRIPTION:
To determine if 600 mg of rifaximin, taken once a day for 14 days by healthy subjects, is safe and effective for the prevention of travellers' diarrhea compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. travelling to Mexico within 72 hours of enrollment
2. read and understand English
3. in good health

Exclusion Criteria:

1. acute diarrhea within previous 7 days
2. taken FQs (any drug in this class), macrolide, azalide, or trimethoprim-sulfamethoxazole within 7 days or enrollment or anytime during study.
3. taken antidiarrheal medication within 24 hours of enrollment or anytime during study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2005-06; Primary Completion 2005-09 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of San Diego, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Derived] Martinez-Sandoval F, Ericsson CD, Jiang ZD, Okhuysen PC, Romero JH, Hernandez N, Forbes WP, Shaw A, Bortey E, DuPont HL. Prevention of travelers' diarrhea with rifaximin in US travelers to Mexico. J Travel Med. 2010 Mar-Apr;17(2):111-7. doi: 10.1111/j.1708-8305.2009.00385.x. PMID 20412178

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm 1: Rifaximin 600 MG QD
- Placebo Arm: Matching Placebo 600MG QD
Period: Overall Study
Arm/Group | Treatment Arm 1 | Placebo Arm
Started | 106 | 104
Completed | 88 | 69
Not Completed | 18 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm 1 | Placebo Arm | Total
Number analyzed (Participants) | 106 | 104 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.5 (9.15) | 22.9 (7.28) | 23.2 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 70 | 136
  Male | 40 | 34 | 74

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Occurrence of Travellers' Diarrhea (TD) for Rifaximin 600 mg QD Compared to Placebo Over 14 Days of Treatment
Description: The efficacy of 14 days of rifaximin 600 mg once daily (QD) compared with placebo when taken by healthy subjects to prevent travelers' diarrhea (TD) resulting from all causes.
Time Frame: 14 days
Population: The Intent to Treat (ITT) population received at least 1 dose of the study drug. For the ITT population, 99 participants were in the rifaximin group and 102 were in the placebo group. The EE consisted of105 of 106 subjects and the placebo group, 100 of 104 subjects were EE. All subject included in Safety analysis
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Arm: Rifaximin
  Rifaximin
- Placebo Arm: Placebo
  Placebo
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 99 | 102
Participants | 15 | 48

ADVERSE EVENTS:
Time Frame: 14 days
Groups:
- Treatment Arm: Rifaximin 600 MG QD
- Placebo: Matching Placebo 600MG QD
Arm/Group | Treatment Arm | Placebo
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/104
Other Adverse Events (participants affected / at risk) | 81/106 | 93/104
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=106) | Placebo (N=104)
Diarrhea (Gastrointestinal disorders) | 62 | 83
Abdominal Pain (Gastrointestinal disorders) | 46 | 63
Defecation Urgency (Gastrointestinal disorders) | 33 | 43
Flatulence (Gastrointestinal disorders) | 27 | 29
Vomiting (Gastrointestinal disorders) | 9 | 8
Rectal tenesmus (Gastrointestinal disorders) | 7 | 13
Hematochezia (Gastrointestinal disorders) | 5 | 6
headache (Nervous system disorders) | 9 | 10
Pyrexia (General disorders) | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes